CLINICAL TRIAL: NCT04295356
Title: A Phase 1, Randomized, Open-label, Two-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics and Safety of the Auto-injector and Pre-filled Syringe of CT-P17 in Healthy Subjects
Brief Title: To Compare the Pharmacokinetics and Safety of the Auto-injector and Pre-filled Syringe of CT-P17
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-P17 1.3
Record Dates: First submitted 2020-03-01; First posted 2020-03-04 (Actual); Results first posted 2020-12-07 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Healthy
MeSH Terms: interventions — CT-P17

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Auto injector (Active Comparator): a single dose (40 mg) of CT-P17 via AI
  Interventions: Biological: CT-P17
- Pre-filled syringe (Active Comparator): a single dose (40 mg) of CT-P17 via PFS
  Interventions: Biological: CT-P17

INTERVENTIONS:
Biological: CT-P17 — subjects will receive a single dose (40 mg) of CT-P17 via AI on Day 1 followed by 10 weeks
  Arms: Auto injector
Biological: CT-P17 — subjects will receive a single dose (40 mg) of CT-P17 via PFS on Day 1 followed by 10 weeks
  Arms: Pre-filled syringe

SUMMARY:
This study was phase 1, randomized, open-label, two-arm, parallel group, single-dose study, which was designed to compare the pharmacokinetics (PK) and safety of CT-P17 SC administration via AI and PFS in healthy subjects. Approximately 180 subjects were enraollend and randomly assigned to one of the two treatment arms in a 1:1 ratio. In each treatment arm, all subjects received a single dose (40 mg) of CT-P17 via either AI or PFS on Day 1 followed by 10 weeks during which PK, safety, and immunogenicity measurements were made. The randomization to treatment assignment was stratified by body weight (≥80 kg vs. <80 kg) as measured on baseline (Day -1), gender (male vs. female) and study center.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria will be considered eligible to participate in the clinical study:

1. Healthy male or female subjects, between the ages of 18 and 55 years, both inclusive (healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and heart rate measurement, 12-lead electrocardiogram [ECG], and clinical laboratory tests prior to the administration of the study drug).
2. Subject with C-reactive protein ≤1.5 times the upper limit of normal (ULN).
3. Subject has adequate liver function as determined by following results:

   * Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5 times ULN and
   * Total bilirubin ≤1.5 times ULN.
4. Subject is informed and able to understand the full nature and purpose of the study, including possible risks and side effects, and is given ample time and opportunity to read and understand this information. The subject has the ability and agrees to cooperate with the investigator and must sign and date the written informed consent prior to performing any of the screening procedures.
5. BMI between 18.0 and 29.9 kg/m2, both inclusive, when rounded to the nearest tenth.
6. Subject and their partner of childbearing potential must agree to use highly effective method of contraception as specified in Section 5.8.2 throughout the study and for 5 months after the administration of the study drug. A man or woman is of childbearing potential if, in the opinion of the investigator, he or she is biologically capable of having children and is sexually active. Male and female subjects and their partners who have been surgically sterilized for less than 24 weeks prior to the date of informed consent must agree to use any medically acceptable methods of contraception. Menopausal females must have experienced their last period more than 1 year prior to the date of informed consent to be classified as not of childbearing potential.

Exclusion Criteria:

Subjects who meet any of the following criteria will not be considered eligible to participate in the clinical study:

1. Subject has a medical history and/or condition including one or more of the following disease(s):

   * History and/or current presence of clinically significant atopy (e.g., allergic asthma, eczematous dermatitis), known or suspected clinically relevant hypersensitivity or allergic reactions to any of the excipients of study drug, other murine and human proteins or immunoglobulin products.
   * History of infection with hepatitis B (active or carrier of hepatitis B), hepatitis C, human immunodeficiency virus (HIV) or syphilis. However, a subject with history of hepatitis B virus is allowed if resolved. Subject will be enrolled based on hepatitis B infection eligibility criteria, specified in Section 6.2.3.
   * History of invasive systemic fungal infections (including histoplasmosis, coccidioidomycosis, candidiasis, aspergillosis, blastomycosis, and pneumocystosis, etc.) or other opportunistic infections judged by the investigator, including local fungal infections or a history of herpes zoster.
   * History of and/or current cardiac (including New York Heart Association class III/IV heart failure), gastrointestinal, renal, endocrine, neurologic, autoimmune, hepatic, hematological (including pancytopenia, aplastic anemia or blood dyscrasia, etc.), metabolic (including diabetes mellitus), or pulmonary disease classed as significant by the investigator.
   * History of any malignancy.
   * History of systemic or local infection, a known risk for developing sepsis, and/or known active inflammatory process or evidence of an infection requiring in-patient hospitalization or intravenous antibiotics within 24 weeks prior to the administration of the study drug (Day 1).
2. Subject is considered to have a significant abnormal cardiac function in investigator's discretion determined by the laboratory results.
3. Subject underwent surgical intervention or an operation within 4 weeks prior to the administration of the study drug (Day 1) or plans to have a surgical procedure during the study period.
4. Subject has active tuberculosis (TB), latent TB (defined as a positive result for interferon-γ release assay [IGRA] with no active lesion in examination of chest X-ray without any sign or symptom of TB), a history of TB, had close contact with a person with active TB or traveled to areas within a high incidence of TB within 8 weeks prior to the administration of the study drug (Day 1) or has plans to travel to the area in which TB is prevalent during the study period. If the result of IGRA is indeterminate at Screening, retest will be allowed only once during the Screening period. If the repeated IGRA result is again indeterminate or positive, the subject will be excluded from the study. If the repeated IGRA result is negative, the subject may be included in the study.
5. Female subject is pregnant or lactating or planning to be pregnant or to breastfeed before, during, or within 5 months after the administration of the study drug (Day 1).
6. Male subject is planning to father a child or donate sperm within 5 months after the administration of the study drug (Day 1).
7. Subject has received tumor necrosis factor-α blockers, or subject who has had exposure of a biologic agent (including but not limited to monoclonal antibodies or fusion protein) within 6 months prior to the administration of the study drug (Day 1).
8. Subject used prescription (excluding hormonal birth control), over-the-counter drugs, dietary supplements, or herbal remedies that could affect the outcome of the study within 2 weeks prior to the administration of the study drug (Day 1).
9. Subject has undergone treatment with an investigational drug or participated in another clinical trial for healthy subject or bioequivalence test within 90 days or 5 half-lives (whichever is longer) prior to the administration of the study drug (Day 1) or plan to do so during the study.
10. Subject received a live or live-attenuated vaccine within 4 weeks prior to the administration of the study drug (Day 1) or plan to do so until the 6 months after Day 1.
11. Subject has donated or lost 450 mL or more of whole blood within 8 weeks, or donated blood components within 4 weeks prior to the administration of the study drug (Day 1).
12. Subject shows reasonable evidence of drug abuse (positive result for drug urine test and/or the opinion of the investigator).
13. Subject has a history or presence of regular consumption exceeding an average weekly intake of >21 units of alcohol in recent 12 weeks prior to the administration of the study drug (Day 1). One unit is equivalent to a half-pint (285 mL) of beer/lager, one measure (25 mL) of spirits, or one small glass (125 mL) of wine. Subject is unwilling to avoid use of alcohol or alcohol containing foods, medications, or beverages within 24 hours prior to admission (Day -1), and each study visit until completion of the study.
14. Subject has smoked 10 or more cigarettes per day in the recent 12 weeks prior to the administration of the study drug (Day 1) and/or is unable to refrain from smoking up to 24 hours after the administration of the study drug.
15. In the opinion of the investigator, the subject is not eligible for the study participation for any reason (including clinical laboratory results) or shows evidence of a condition (e.g., psychological or emotional problem, any disorder or resultant therapy) that is likely to invalidate an informed consent or limit the ability of the subject to comply with the protocol requirements. Subject is unable to understand the protocol requirements, instructions, study-related restrictions, or the nature, scope, and possible consequences of the clinical study or is unable to give written informed consent or to comply fully with the protocol.
16. Subject is vulnerable (e.g., employees of the study center or any other individuals involved with the conduct of the study, or immediate family members of such individuals, persons kept in prison, or other institutionalized persons by law enforcement).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Hyun Kim, Dr, Study Director — Celltrion
Locations (1):
- PPD Development, LP, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Davidson A, Brimhall D, Kay J, Keystone E, Lee SJ, Kim SH, Bae YJ, Choi EJ, Furst DE. Randomised, phase I pharmacokinetic study of adalimumab biosimilar CT-P17 (40 mg/0.4 mL) by autoinjector and prefilled syringe in healthy subjects. Br J Clin Pharmacol. 2021 Nov;87(11):4323-4333. doi: 10.1111/bcp.14850. Epub 2021 May 9. PMID 33822406

RESULTS

PARTICIPANT FLOW:
Groups:
- Auto Injector: a single dose (40 mg) of CT-P17 via AI
  CT-P17: all subjects will receive a single dose (40 mg) of CT-P17 via either AI or PFS on Day 1 followed by 10 weeks
- Pre-filled Syringe: a single dose (40 mg) of CT-P17 via PFS
  CT-P17: all subjects will receive a single dose (40 mg) of CT-P17 via either AI or PFS on Day 1 followed by 10 weeks
Period: Overall Study
Arm/Group | Auto Injector | Pre-filled Syringe
Started | 93 | 87
Completed | 92 | 83
Not Completed | 1 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 3
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Auto Injector | Pre-filled Syringe | Total
Number analyzed (Participants) | 93 | 87 | 180
Age, Continuous [Mean (Full Range); unit: years] | 35.2 [18 to 55] | 36.7 [18 to 55] | 35.9 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 90
  Male | 48 | 42 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 25 | 57
  Not Hispanic or Latino | 61 | 62 | 123
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 39 | 73
  White | 53 | 47 | 100
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 93 | 87 | 180
Female fertility status [Count of Participants; unit: Participants]
  Surgically sterilized | 10 | 9 | 19
  Post-menopausal | 3 | 0 | 3
  Potentially able to bear children | 32 | 36 | 68
  Not applicable (male) | 48 | 42 | 90
Screening height [Mean (Standard Deviation); unit: cm] | 168.35 (9.266) | 169.57 (9.795) | 168.94 (9.518)
Screening weight [Mean (Standard Deviation); unit: kg] | 71.61 (12.888) | 73.12 (12.574) | 72.34 (12.725)
Screening BMI [Mean (Standard Deviation); unit: kg/m2] | 25.12 (3.029) | 25.32 (2.947) | 25.22 (2.983)
Day -1 BMI [Mean (Standard Deviation); unit: kg/m2] | 25.26 (2.967) | 25.50 (2.939) | 25.38 (2.948)
Day -1 weight category [Count of Participants; unit: Participants]
  Weight <80 kg | 65 | 62 | 127
  Weight ≥80 kg | 28 | 25 | 53

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration (Cmax)
Description: To demonstrate the PK similarity of CT-P17 SC administration via AI versus PFS in healthy subjects
Time Frame: Day 1 predose, 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504 hours, Days 29, 43, 57, 71 postdose
Population: Pharmacokinetics population
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Auto Injector | Pre-filled Syringe
Number analyzed (Participants) | 84 | 76
μg/mL | 4.141 (1.5479) | 3.908 (1.2620)
Statistical Analysis 1: Comparison: Auto Injector vs Pre-filled Syringe; Equivalence test in Cmax between CT-P17 AI and CT-P17 PFS; Test type: Equivalence — The 90% confidence interval of the ratio of geometric least squares means of Cmax was estimated to assess the PK similarity between CT-P17 AI and CT-P17 PFS (bioequivalence margin of 80% to 125%); ANCOVA; The stratification factors (gender [male or female], study center, and body weight as measured on Day -1) were included in ANCOVA model as covariates; Ratio of geometric least squares means = 102.60, 90% CI 2-sided [94.08 to 111.90]

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC0-inf)
Description: To demonstrate the PK similarity of CT-P17 SC administration via AI versus PFS in healthy subjects
Time Frame: Day 1 predose, 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504 hours, Days 29, 43, 57, 71 postdose
Population: Pharmacokinetics population; AUC0-inf PK parameter values were excluded from the statistical analysis after not meeting 1 or more of the following criteria; terminal elimination rate constant was calculated with an adjusted correlation coefficient r2 of ≥0.85 and/or a %AUCextrap (percentage of the area extrapolated for calculation of area under the concentration-time curve from time zero to infinity) ≤20%.
Measure: Mean (Standard Deviation); unit: h•μg/mL
Arm/Group | Auto Injector | Pre-filled Syringe
Number analyzed (Participants) | 69 | 63
h•μg/mL | 2819.5 (945.82) | 2684.5 (1031.16)
Statistical Analysis 1: Comparison: Auto Injector vs Pre-filled Syringe; Equivalence test in AUC0-inf between CT-P17 AI and CT-P17 PFS; Test type: Equivalence — The 90% confidence interval of the ratio of geometric least squares means of AUC0-inf was estimated to assess the PK similarity between CT-P17 AI and CT-P17 PFS (bioequivalence margin of 80% to 125%); ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric least squares means = 103.64, 90% CI 2-sided [93.98 to 114.29]

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Zero to the Last Quantifiable Concentration (AUC0-last))
Description: To demonstrate the PK similarity of CT-P17 SC administration via AI versus PFS in healthy subjects
Time Frame: Day 1 predose, 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504 hours, Days 29, 43, 57, 71 postdose
Population: Pharmacokinetics population
Measure: Mean (Standard Deviation); unit: h•μg/mL
Arm/Group | Auto Injector | Pre-filled Syringe
Number analyzed (Participants) | 84 | 76
h•μg/mL | 2451.3 (1086.28) | 2292.9 (1026.99)
Statistical Analysis 1: Comparison: Auto Injector vs Pre-filled Syringe; Equivalence test in AUC0-last between CT-P17 AI and CT-P17 PFS; Test type: Equivalence — The 90% confidence interval of the ratio of geometric least squares means of AUC0-last was estimated to assess the PK similarity between CT-P17 AI and CT-P17 PFS (bioequivalence margin of 80% to 125%); ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric least squares means = 105.36, 90% CI 2-sided [91.09 to 121.86]

4. Secondary Outcome: Time to Maximum Serum Concentration (Tmax)
Description: To evaluate the additional PK parameters of CT-P17 SC administration via AI versus PFS in healthy subjects
Time Frame: Day 1 predose, 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504 hours, Days 29, 43, 57, 71 postdose
Population: Pharmacokinetics population
Measure: Median (Full Range); unit: hour
Arm/Group | Auto Injector | Pre-filled Syringe
Number analyzed (Participants) | 84 | 76
hour | 132 [24.00 to 504.18] | 132 [48.00 to 505.97]

5. Secondary Outcome: Terminal Elimination Half-life (t1/2)
Description: To evaluate the additional PK parameters of CT-P17 SC administration via AI versus PFS in healthy subjects
Time Frame: Day 1 predose, 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504 hours, Days 29, 43, 57, 71 postdose
Population: Pharmacokinetics population; t1/2 PK parameter values were excluded from the statistical analysis after not meeting 1 or more of the following criteria; terminal elimination rate constant was calculated with an adjusted correlation coefficient r2 of ≥0.85 and/or a %AUCextrap (percentage of the area extrapolated for calculation of area under the concentration-time curve from time zero to infinity) ≤20%.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Auto Injector | Pre-filled Syringe
Number analyzed (Participants) | 69 | 63
hour | 369.0 (139.76) | 355.4 (141.80)

6. Secondary Outcome: Terminal Elimination Rate Constant (λz)
Description: To evaluate the additional PK parameters of CT-P17 SC administration via AI versus PFS in healthy subjects
Time Frame: Day 1 predose, 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504 hours, Days 29, 43, 57, 71 postdose
Population: Pharmacokinetics population; λz PK parameter values were excluded from the statistical analysis after not meeting 1 or more of the following criteria; terminal elimination rate constant was calculated with an adjusted correlation coefficient r2 of ≥0.85 and/or a %AUCextrap (percentage of the area extrapolated for calculation of area under the concentration-time curve from time zero to infinity) ≤20%.
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Auto Injector | Pre-filled Syringe
Number analyzed (Participants) | 69 | 63
1/h | 0.0022 (0.00110) | 0.0023 (0.00100)

7. Secondary Outcome: Apparent Total Body Clearance (CL/F)
Description: To evaluate the additional PK parameters of CT-P17 SC administration via AI versus PFS in healthy subjects
Time Frame: Day 1 predose, 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504 hours, Days 29, 43, 57, 71 postdose
Population: Pharmacokinetics population; CL/F PK parameter values were excluded from the statistical analysis after not meeting 1 or more of the following criteria; terminal elimination rate constant was calculated with an adjusted correlation coefficient r2 of ≥0.85 and/or a %AUCextrap (percentage of the area extrapolated for calculation of area under the concentration-time curve from time zero to infinity) ≤20%.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Auto Injector | Pre-filled Syringe
Number analyzed (Participants) | 69 | 63
L/h | 0.016 (0.00740) | 0.017 (0.00599)

8. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase After Non-IV Administration (Vz/F)
Description: To evaluate the additional PK parameters of CT-P17 SC administration via AI versus PFS in healthy subjects
Time Frame: Day 1 predose, 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504 hours, Days 29, 43, 57, 71 postdose
Population: Pharmacokinetics population; Vz/F PK parameter values were excluded from the statistical analysis after not meeting 1 or more of the following criteria; terminal elimination rate constant was calculated with an adjusted correlation coefficient r2 of ≥0.85 and/or a %AUCextrap (percentage of the area extrapolated for calculation of area under the concentration-time curve from time zero to infinity) ≤20%.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Auto Injector | Pre-filled Syringe
Number analyzed (Participants) | 69 | 63
L | 7.9 (2.75) | 7.9 (2.71)

9. Secondary Outcome: Percentage of the Area Extrapolated for Calculation of AUC0-inf (%AUCextrap)
Description: To evaluate the additional PK parameters of CT-P17 SC administration via AI versus PFS in healthy subjects
Time Frame: Day 1 predose, 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 192, 336, 504 hours, Days 29, 43, 57, 71 postdose
Population: Pharmacokinetics population; %AUCextrap PK parameter values were excluded from the statistical analysis after not meeting 1 or more of the following criteria; terminal elimination rate constant was calculated with an adjusted correlation coefficient r2 of ≥0.85 and/or a %AUCextrap (percentage of the area extrapolated for calculation of area under the concentration-time curve from time zero to infinity) ≤20%.
Measure: Mean (Standard Deviation); unit: % of AUCextrap
Arm/Group | Auto Injector | Pre-filled Syringe
Number analyzed (Participants) | 69 | 63
% of AUCextrap | 7.3 (4.52) | 7.1 (4.52)

10. Secondary Outcome: Summary of Immunogenicity Assay
Description: To evaluate immunogenicity of CT-P17 SC administration via AI versus PFS in healthy subjects
Time Frame: Day 1 predose, Days 15, 29, 57, 71 postdose
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Auto Injector | Pre-filled Syringe
Number analyzed (Participants) | 93 | 87
Participants
  Baseline (Day 1 predose) ADA: Positive | 10 | 5
  Baseline (Day 1 predose) ADA: Negative | 83 | 82
  Baseline (Day 1 predose) ADA: Missing or not applicable | 0 | 0
  Day 15 ADA: Positive | 62 | 59
  Day 15 ADA: Negative | 30 | 27
  Day 15 ADA: Missing or not applicable | 1 | 1
  Day 29 ADA: Positive | 78 | 73
  Day 29 ADA: Negative | 10 | 11
  Day 29 ADA: Missing or not applicable | 5 | 3
  Day 57 ADA: Positive | 82 | 73
  Day 57 ADA: Negative | 6 | 7
  Day 57 ADA: Missing or not applicable | 5 | 7
  End-of-study ADA: Positive | 87 | 78
  End-of-study ADA: Negative | 4 | 6
  End-of-study ADA: Missing or not applicable | 2 | 3
  Baseline (Day 1 predose) NAb: Positive | 0 | 0
  Baseline (Day 1 predose) NAb: Negative | 10 | 5
  Baseline (Day 1 predose) NAb: Missing or not applicable | 83 | 82
  Day 15 NAb: Positive | 21 | 25
  Day 15 NAb: Negative | 41 | 34
  Day 15 NAb: Missing or not applicable | 31 | 28
  Day 29 NAb: Positive | 39 | 44
  Day 29 NAb: Negative | 39 | 29
  Day 29 NAb: Missing or not applicable | 15 | 14
  Day 57 NAb: Positive | 65 | 60
  Day 57 NAb: Negative | 17 | 13
  Day 57 NAb: Missing or not applicable | 11 | 14
  End-of-study NAb: Positive | 73 | 68
  End-of-study NAb: Negative | 14 | 10
  End-of-study NAb: Missing or not applicable | 6 | 9

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Auto Injector | Pre-filled Syringe
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/87
Serious Adverse Events (participants affected / at risk) | 2/93 | 0/87
Other Adverse Events (participants affected / at risk) | 55/93 | 45/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Auto Injector (N=93) | Pre-filled Syringe (N=87)
Viral meningitis (Infections and infestations) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Auto Injector (N=93) | Pre-filled Syringe (N=87)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Eyelid irritation (Eye disorders) | 0 | 2
Vision blurred (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3
Toothache (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Chills (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 2
Feeling hot (General disorders) | 1 | 0
Injection site reaction (General disorders) | 8 | 6
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 3 | 1
Cystitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Pyuria (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 3 | 2
Vaginal infection (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 2 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 3
Blood creatine phosphokinase MB increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 7 | 4
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 5 | 5
Electrocardiogram T-wave abnormal (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 1
Urine output decreased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 8 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Aura (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 11 | 8
Paraesthesia (Nervous system disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT04295356/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT04295356/SAP_001.pdf